CLINICAL TRIAL: NCT04757909
Title: Early Detection of Anemizations in Primary Care Using Hemoglobinometer: Randomized Clinical Trial Protocol.
Brief Title: Detection of Anemizations in Primary Care.
Acronym: ANHEMOG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 4R17/013; 4R18/08 (Other Grant/Funding Number: Academia de Ciencias Médicas filial de Maresme); 4R17/013 (Other Grant/Funding Number: Direcció Atenció Primària Metropolitana Nord)
Record Dates: First submitted 2021-02-15; First posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Anemia; Red Blood Cell Transfusion
Keywords: Haemoglobinometry; Primary Care Nursing,; Advanced Practice Nursing
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monthly Haemoglobinometry (Experimental)
  Interventions: Diagnostic Test: Monthly Haemoglobinometry
- Routine monitoring (No Intervention)

INTERVENTIONS:
Diagnostic Test: Monthly Haemoglobinometry — Monthly measurement of capillary hemoglobin with non-invasive techniques in primary health care.
  Inclusion in a transfusion circuit with referral to a hospital day hospital if necessary.
  Arms: Monthly Haemoglobinometry

SUMMARY:
Objective: To evaluate the effect of the use of the hemoglobinometer in primary care on the clinical results of patients with chronic anemia.

Methods: The ANHEMOG study is a randomized controlled trial with two parallel arms, intervention and control. It was approved at december 11, 2017. The study randomizes 138 patients with chronic anemia. In the intervention arm, a monthly capillary hemoglobin measurement will be performed with a hemoglobinometer. If a decrease in hemoglobin concentration is detected, an existing transfusion circuit will be followed. Social, demographic and quality of life variables will be collected from all participants.

Hypothesis:

The results of the research will have an impact on people with chronic anemia who would receive red blood cell transfusion when needed without delay. The improvement in the times of action would reduce decompensations from chronic diseases, visits to the emergency room and hospital admissions, and therefore would improve the quality of life of these patients. Furthermore, the management of the different interventions by the Case Management Nurse (EGC), in this regard, improves the current fragmentation of the different levels of care.

ELIGIBILITY:
Inclusion Criteria:

* People over 40 years old
* Had received 2 or more red blood cell transfusions due to chronic disease, during a year.
* The health provider in Primary Care is the Institut Català de la Salut.

Exclusion Criteria:

* Presenting kidney failure on hemodialysis treatment.
* Being in palliative care situation
* Presenting a moderate-severe cognitive impairment, with a Pfeiffer scale score higher than 5.
* Not having a caregiver able to detect signs of decompensation.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2017-03-30 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Mean Number of hospital admissions | 6 and 12 months.
  Anual mean of hospital admissions caused by haemoglobin concentration decline.
Mean Number of visits to the emergency room | 6 and 12 months.
  Anual mean of visits to the emergency room caused by haemoglobin concentration decline.

SECONDARY OUTCOMES:
Quality of life self-assessment. | 6 and 12 months.
  WHOQOL-BREF questionnaire.
Satisfaction with the intervention. | 6 and 12 months.
  Ad-hoc questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- CAP La Llàntia, Mataró, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Study protocol will be sent to publication in the next months
Supporting Information: Study Protocol
Time Frame: Open access to read as soon as published
Access Criteria: Open

REFERENCES:
- [Derived] Radford M, Estcourt LJ, Sirotich E, Pitre T, Britto J, Watson M, Brunskill SJ, Fergusson DA, Doree C, Arnold DM. Restrictive versus liberal red blood cell transfusion strategies for people with haematological malignancies treated with intensive chemotherapy or radiotherapy, or both, with or without haematopoietic stem cell support. Cochrane Database Syst Rev. 2024 May 23;5(5):CD011305. doi: 10.1002/14651858.CD011305.pub3. PMID 38780066
- [Derived] Luengo BT, Garcia-Sierra R, Trinxant MAW, Mondelo ED, Baseda RM, Blanch MML, Del Pilar Montero Alia M, Toran-Monserrat P. Early detection of anaemia in primary care with haemoglobinometry: ANHEMOG clinical trial protocol. BMC Fam Pract. 2021 Oct 8;22(1):199. doi: 10.1186/s12875-021-01548-z. PMID 34625027